CLINICAL TRIAL: NCT00857805
Title: Randomized Controlled Trial of Transarterial Chemoembolization Versus Proton Beam Radiotherapy for the Treatment of Hepatocellular Carcinoma
Brief Title: Transarterial Chemoembolization Versus Proton Beam Radiotherapy for the Treatment of Hepatocellular Carcinoma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Loma Linda University (Other)
Responsible Party: Principal Investigator, David Bush, Medical Doctor, Loma Linda University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 58348
Record Dates: First submitted 2009-03-05; First posted 2009-03-09 (Estimated); Results first posted 2024-05-31 (Actual); Last update posted 2024-05-31 (Actual); Status verified 2024-05

CONDITIONS: Carcinoma, Hepatocellular
Keywords: Transarterial chemoembolization; Carcinoma, Hepatocellular; Proton Beam Radiotherapy
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Chlorotrianisene

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Transarterial Chemoembolization (Active Comparator): Transarterial Chemoembolization
  Interventions: Procedure: Transarterial Chemoembolization
- Proton Beam Radiotherapy (Active Comparator): Proton Beam Radiotherapy
  Interventions: Radiation: Proton Beam Radiotherapy

INTERVENTIONS:
Procedure: Transarterial Chemoembolization — Application of carboplatin, doxorubicin in ethiodol into the artery for one or more sessions.
  Other Names: (TACE)
  Arms: Transarterial Chemoembolization
Radiation: Proton Beam Radiotherapy — Fifteen consecutive sessions
  Arms: Proton Beam Radiotherapy

SUMMARY:
Patients with liver tumor burden that exceeds Milan criteria are considered to receive one of the following locoregional treatments: transarterial chemoembolization (TACE), radiofrequency ablation (RFA), percutaneous ethanol injection and proton beam radiation (PBR). The goals of these treatments are to control tumor growth, to downstage tumor size to meet Milan criteria, and to improve survival. Patients who exceed the Milan criteria benefit from tumor downstaging as a result of treatment. Patients who meet Milan criteria benefit from tumor control to bridge them to liver transplantation. TACE is considered the most common locoregional treatment that is used to treat hepatocellular carcinoma (HCC). Proton beam radiotherapy has been used in treating HCC in a few centers across the globe. Phase I and II trials showed a satisfactory safety and efficacy results. Loma Linda University Medical Center is one of these pioneering centers that use proton beam as a treatment for HCC. This is the first randomized trial in the medical field that will compare head-to-head the efficacy of TACE versus proton beam in treating HCC patients.

ELIGIBILITY:
Inclusion Criteria:

1. Patients are candidates to receive both proton beam and TACE
2. Patients with no evidence of metastasis or macrovascular invasion
3. Patients with tumor burden that meets San Francisco criteria

Exclusion Criteria:

1. Patients who are candidates for surgical resection
2. Patients with lesion < 2 cm
3. Patients who have contraindication to receive either TACE or proton
4. Patients with serum alpha fetoprotein > 500
5. Patients with metastasis or macrovascular invasion
6. Patients treated previously for HCC by any locoregional treatment
7. Patients with prior liver transplant
8. Patients with Child class C
9. Patients with MELD score of > 25
10. Patients with other comorbid diseases that may impact survival
11. Patients with ongoing alcohol intake
12. Patients with active sepsis
13. Patients with gastrointestinal bleeding within a week
14. Patients unwilling to sign informed consent form
15. Patients with history of noncompliance

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2009-01-07 (Actual); Primary Completion 2021-07-07 (Actual); Study Completion 2021-07-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael deVera, MD, Principal Investigator — Loma Linda University Medical Center
Locations (1):
- Loma Linda University Medical Center, Loma Linda, California, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Transarterial Chemoembolization | Proton Beam Radiotherapy
Started | 40 | 36
Completed | 39 | 35
Not Completed | 1 | 1
Not completed — Withdrawal by Subject | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Transarterial Chemoembolization | Proton Beam Radiotherapy | Total
Number analyzed (Participants) | 39 | 35 | 74
Age, Customized [Mean (Standard Deviation); unit: years] | 59.6 (9.15) | 61.7 (8.51) | 60.65 (8.83)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 8 | 21
  Male | 26 | 27 | 53
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 39 | 35 | 74

OUTCOME MEASURES:

1. Primary Outcome: Two Year Overall Survival
Description: Comparison between arms of the percentage of patient alive 2 years following study treatment.
Time Frame: 24 Months
Population: Eligible subjects were adult patients with newly diagnosed and previously untreated HCC. All subjects had characteristic findings of HCC on contrast-enhanced magnetic resonance imaging (MRI) and/or computed tomography (CT) scanning or histologic proof with biopsy. Patients were required to have tumors that were within the Milan or San Francisco criteria, although eligibility for transplant was not required.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Transarterial Chemoembolization | Proton Beam Radiotherapy
Number analyzed (Participants) | 39 | 35
percentage of participants | 65 [52 to 83] | 68 [54 to 86]

ADVERSE EVENTS:
Time Frame: 30 months
Description: 74 participants at risk
Arm/Group | Transarterial Chemoembolization | Proton Beam Radiotherapy
All-Cause Mortality (participants affected / at risk) | 13/39 | 16/35
Serious Adverse Events (participants affected / at risk) | 8/39 | 2/35
Other Adverse Events (participants affected / at risk) | 39/39 | 35/35
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Transarterial Chemoembolization (N=39) | Proton Beam Radiotherapy (N=35)
Liver Failure (Gastrointestinal disorders) | 8 (8) | 2 (2)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Transarterial Chemoembolization (N=39) | Proton Beam Radiotherapy (N=35)
Abdominal Pain (Hepatobiliary disorders) | 23 | 7
Nausea (Gastrointestinal disorders) | 10 | 9
Vomiting (Gastrointestinal disorders) | 6 | 0
Diarrhea (Gastrointestinal disorders) | 1 | 3
GI Ulcer (Gastrointestinal disorders) | 0 | 1
GI Bleed (Gastrointestinal disorders) | 2 | 2
Erythema (Skin and subcutaneous tissue disorders) | 0 | 12
Fatigue (General disorders) | 4 | 11

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2009-03-05): https://cdn.clinicaltrials.gov/large-docs/05/NCT00857805/Prot_SAP_000.pdf